CLINICAL TRIAL: NCT00533039
Title: sPLA2 Inhibition to Decrease Enzyme Release After PCI (SPIDER-PCI) Trial
Brief Title: sPLA2 Inhibition to Decrease Enzyme Release After PCI Trial
Acronym: SPIDER-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Anthera Pharmaceuticals (Industry)
Responsible Party: Vladimir Dzavik, MD, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPIDER001; A Sub-study of SPIDER-PCI
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — varespladib; varespladib methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Subjects take 2 tablets BID. Placebo tablets are identical to active medication.
  Interventions: Drug: placebo
- Varespladib (A-002) (Experimental): Subjects take 250mg tablets BID beginning 3-5 days pre-angioplasty and for 5 days post-angioplasty.
  Interventions: Drug: Varespladib (A-002)

INTERVENTIONS:
Drug: Varespladib (A-002) — 250mg tablets BID for 3-5 days pre-angioplasty and 5 days post-angioplasty.
  Arms: Varespladib (A-002)
Drug: placebo — 250mg tablets BID 3-5 days pre-angioplasty and 5 days post-angioplasty.
  Arms: Control

SUMMARY:
As evidence accumulates that atherogenesis or Coronary Artery Disease (CAD) may not be simply a disorder of lipid metabolism, but an inflammatory disease, the focus of treatment has shifted. A-002 or Varespladib is an anti-inflammatory drug for treatment of chronic and acute diseases. It acts by inhibiting secretory phospholipase A2 (sPLA2 ) - one of a family of enzymes leading to inflammation - which may be important in: 1) the development of atherosclerosis and 2) the increase in occurence of cardiovascular events after angioplasty. Previous studies have demonstrated that sPLA2: 1) facilitates the pro-atherogenic effects of low-density (LDL or bad cholesterol) and 2) increased levels post-angioplasty correlate with an increased risk of events at followup contact. Therefore this study proposes to investigate the ability of A-002 to prevent or reduce myocardial damage after angioplasty by inhibiting the cascade of inflammatory mediators.

Substudy - Subjects who agree will also have a vascular ultrasound 24h post-PCI to assess endothelial function.

DETAILED DESCRIPTION:
Tissue injury after angioplasty is likely due to micro-emboli from mechanical trauma to a thrombotic lesion during angioplasty. In response to the ischemia sPLA2, possibly localized within atherosclerotic vascular tissue as well as from macrophages and monocytes, is released. Following ischemia-induced release, sPLA2 can bind to ischemically challenged cardiomyocytes and adversely affect their survival either directly through toxic effects on cardiomyocytes or indirectly by facilitating inflammation. It may be possible through sPLA2 inhibition to salvage non-lethally jeopardized cells following an ischemic episode thereby reducing the infarcted area and amount of tissue damage. Previous studies in patients with unstable angina support this hypothesis, and conclude that sPLA2 levels can be used to predict clinical outcomes. We hypothesize that sPLA2 inhibition with A-002 will reduce myocardial injury post-angioplasty.

Substudy - Peripheral vascular ultrasound should be done prior to receiving study drug and 24h post-PCI. Coronary endothelial function will be assessed at the time of PCI.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age undergoing elective PCI, with or without stenting

Exclusion Criteria:

* ST elevation MI or any troponin elevation (non-STEMI) within preceding 10days
* Elevation of CK-MB or troponin I at baseline
* Recent (4 weeks) coronary bypass surgery
* NYHA class III-IV heart failure
* Left ventricular ejection fraction < 0.30
* Severe valvular heart disease
* Chronic inflammatory disease (e.g., lupus, rheumatoid arthritis, inflammatory bowel disease), or patients receiving steroid drugs
* Presence of severe liver disease with cirrhosis
* Recent active hepatitis
* Active chronic hepatitis
* ALT or AST > 3 × upper limit of normal (ULN)
* Biliary obstruction with hyperbilirubinemia (total bilirubin > 2 × ULN)
* Moderate or severe renal impairment (creatinine > 1.5 × ULN)
* Nephrotic syndrome or subjects undergoing dialysis
* Uncontrolled diabetes (HbA1c > 11% 1 month prior to screening)
* Initiation of statin therapy within 30 days
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be incidence of myocardial injury as evidenced by elevation of CK-MB or troponin I above the upper limit of normal. | 8 hours and 18-24 hours post-angioplasty

SECONDARY OUTCOMES:
A secondary endpoint will be occurrence of elevation of CK-MB or troponin I above the upper limit of normal. | 8 and 18-24 hours post-angioplasty
A secondary endpoint will be occurrence of any major adverse cardiac events (MACE). | 30 days post-angioplasty
A secondary outcome will be serum sPLA2 activity. | 5-7 days post-angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, Study Chair — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dzavik V, Lavi S, Thorpe K, Yip PM, Plante S, Ing D, Overgaard CB, Osten MD, Lan J, Robbins K, Miner SE, Horlick EM, Cantor WJ. The sPLA2 Inhibition to Decrease Enzyme Release after Percutaneous Coronary Intervention (SPIDER-PCI) trial. Circulation. 2010 Dec 7;122(23):2411-8. doi: 10.1161/CIRCULATIONAHA.110.950733. Epub 2010 Nov 22. PMID 21098449